CLINICAL TRIAL: NCT00692276
Title: A Prospective, Multi-Center, Randomized Study Comparing the VertiFlex® Superion™ Interspinous Spacer (ISS) to the X-STOP® Interspinous Process Decompression (IPD®) System in Patients With Moderate Lumbar Spinal Stenosis
Brief Title: Investigating Superion™ In Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: VertiFlex, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-VISS-01
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Lumbar Spinal Stenosis; Intermittent Claudication
MeSH Terms: conditions — Spinal Stenosis; Intermittent Claudication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Interspinous Process Spacer Device
  Interventions: Device: Superion™ Interspinous Spacer
- 2 (Active Comparator): Interspinous Process Spacer Device
  Interventions: Device: X-STOP® IPD® Device

INTERVENTIONS:
Device: Superion™ Interspinous Spacer — Implantation of interspinous process spacer to treat lumbar spinal stenosis
  Arms: 1
Device: X-STOP® IPD® Device — Implantation of interspinous process spacer to treat lumbar spinal stenosis
  Arms: 2

SUMMARY:
The proposed prospective, multi-center, randomized clinical trial is designed to evaluate the safety and effectiveness of the Superion™ ISS compared to the X-STOP® IPD® device in healthy adults suffering from at least 6 months of moderate spinal stenosis symptoms who have been unresponsive to conservative care.

DETAILED DESCRIPTION:
The proposed prospective, multi-center, randomized clinical trial is designed to evaluate the safety and effectiveness of the Superion™ ISS compared to the X-STOP® IPD® device in healthy adults suffering from at least 6 months of moderate spinal stenosis symptoms who have been unresponsive to conservative care. The study endpoint is the rate of overall subject success at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 45 years of age
* Persistent leg/buttock/groin pain, with or without back pain, that is relieved by flexion activities (example: sitting or bending over a shopping cart)
* Diagnosis of degenerative spinal stenosis of the lumbar spine, defined as the narrowing of the midline sagittal spinal canal (central) and/or narrowing between the facet superior articulating process (SAP), the posterior vertebral margin (lateral recess), and the nerve root canal (foraminal)
* Must be able to sit for 50 minutes without pain and to walk 50 feet or more

Exclusion Criteria:

* Axial back pain only
* Fixed motor deficit
* Diagnosis of lumbar spinal stenosis which requires any direct neural decompression or surgical intervention other than those required to implant the control or experimental device
* Unremitting pain in any spinal position
* Significant peripheral neuropathy or acute denervation secondary to radiculopathy
* Lumbar spinal stenosis at more than two levels determined pre-operatively to require surgical intervention
* Significant instability of the lumbar spine as defined by 3mm translation or 5 degrees angulation
* Sustained pathologic fractures of the vertebrae or multiple fractures of the vertebrae and/or hips
* Spondylolisthesis or degenerative spondylolisthesis greater than grade 1.0 (on a scale of 1 to 4)
* Spondylolysis (pars fracture)
* Morbid obesity, defined as Body Mass Index (BMI) greater than 40kg/m2
* Insulin-dependent diabetes mellitus
* Prior surgery of the lumbar spine
* Cauda equina syndrome (defined as neural compression causing neurogenic bowel or bladder dysfunction)
* Infection in the disc or spine, past or present
* Paget's disease at involved segment or metastasis to the vertebra, osteomalacia, or other metabolic bone disease
* Tumor in the spine or a malignant tumor except for basal cell carcinoma
* Involved in pending litigation of the spine or worker's compensation related to the back

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2008-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — Boston Scientific Corporation
Locations (32):
- United States (32):
  - Arizona Center for Neurosurgery, Phoenix, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - D.I.S.C. Sports and Spine Center, Beverly Hills, California
  - Tower Orthopaedics and Sports Medicine/ Institute for Advanced Spinal Research, Beverly Hills, California
  - Orange County Neurosurgical Associates, Laguna Hills, California
  - Brain and Spine Research Institute, Los Angeles, California
  - Pacific Pain Medicine Consultants/Pacific Surgery Center, Oceanside, California
  - University of Colorado Hospital- The Spine Center- Anshutz Outpatient Pavilion, Aurora, Colorado
  - Durango Orthopedic Associates, P.C./Spine Colorado, Durango, Colorado
  - Colorado Spine And Scoliosis Institute, Littleton, Colorado
  - Yale University, New Haven, Connecticut
  - The George Washington Universtiy Medical Facility, Washington D.C., District of Columbia
  - Florida Research Associates, LLC, DeLand, Florida
  - Shrock Orthopedic Research, Fort Lauderdale, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Greater Baltimore Neurosurgical Associates at GBMA, Baltimore, Maryland
  - Sports Medicine North, Peabody, Massachusetts
  - Institute for Low Back and Neck Care, Minneapolis, Minnesota
  - Orthopedics Associates of the Greater Lehigh Valley, Phillipsburg, New Jersey
  - Spine Care and Rehabilitation, Inc., Roseland, New Jersey
  - Stony Brook University Medical Center, Dept. of Neurological Surgery, Stony Brook, New York
  - Upstate Medical Universtiy-Department of Orthopedics- Institute for Spine Care, Syracuse, New York
  - Triangle Orthopaedic Associates, Durham, North Carolina
  - NeuroSpine Institute, LLC, Eugene, Oregon
  - Performance Spine and Sports Physicians, Pottstown, Pennsylvania
  - OrthopaediCare (Abington Orthopaedic Specialists), Willow Grove, Pennsylvania
  - New England Center for Clinical Research, Cranston, Rhode Island
  - East Tennessee Brain & Spine Center, Johnson City, Tennessee
  - Texas Back Institute, Plano, Texas
  - Orthopedics International Spine, Seattle, Washington
  - The Center for Pain Relief, Inc, Charleston, West Virginia

REFERENCES:
- [Derived] Patel VV, Whang PG, Haley TR, Bradley WD, Nunley PD, Miller LE, Block JE, Geisler FH. Two-year clinical outcomes of a multicenter randomized controlled trial comparing two interspinous spacers for treatment of moderate lumbar spinal stenosis. BMC Musculoskelet Disord. 2014 Jul 5;15:221. doi: 10.1186/1471-2474-15-221. PMID 24996648
- [Derived] Loguidice V, Bini W, Shabat S, Miller LE, Block JE. Rationale, design and clinical performance of the Superion(R) Interspinous Spacer: a minimally invasive implant for treatment of lumbar spinal stenosis. Expert Rev Med Devices. 2011 Jul;8(4):419-26. doi: 10.1586/erd.11.24. PMID 21728727

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 - Study Treatment: Interspinous Process Spacer Device
  Superion™ Interspinous Spacer: Implantation of interspinous process spacer to treat lumbar spinal stenosis
- 2 - Active Control Treatment: Interspinous Process Spacer Device
  X-STOP® IPD® Device: Implantation of interspinous process spacer to treat lumbar spinal stenosis
Period: Randomized Population
Arm/Group | 1 - Study Treatment | 2 - Active Control Treatment
Started | 190 | 201
Completed | 190 | 201
Not Completed | 0 | 0
Period: Completed 24 Months
Arm/Group | 1 - Study Treatment | 2 - Active Control Treatment
Started | 190 | 201
Completed | 183 | 187
Not Completed | 7 | 14

BASELINE CHARACTERISTICS:
Groups:
- 1 - Study Treatment: Superion™ Interspinous Spacer
- 2 - Active Control Treatment: X-STOP® IPD® Device
- Total: Total of all reporting groups
Arm/Group | 1 - Study Treatment | 2 - Active Control Treatment | Total
Number analyzed (Participants) | 190 | 201 | 391
Age, Customized [Mean (Standard Deviation); unit: years] | 66.9 (9.4) | 66.2 (10.2) | 66.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 72 | 152
  Male | 110 | 129 | 239
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 11 | 16
  Not Hispanic or Latino | 185 | 190 | 375
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Clinically Significant Improvement in Outcomes
Description: Where clinically significant improvement in outcomes compared to baseline, as determined by meeting the following:
  * At least two of three domains of the Zurich Claudication Questionnaire (ZCQ) [validated, condition-specific patient-reported questionnaire that captures data in three distinct domains]
    * Improvement in physical function by ≥0.5 points
    * Improvement in symptom severity by ≥0.5 points
    * "Satisfied" or "somewhat satisfied" as defined by a score of ≤ 2.5 points on the patient satisfaction domain
  * No re-operations, revisions, removals or supplemental fixation at the index level(s)
  * No major implant- or procedure-related complications:
    * No dislodgement, migration, or deformation
    * No new or persistent worsened neurological deficit at the index level
    * No spinous process fractures
    * No deep infection, death, or other permanent device attributed disability
  * No clinically significant confounding treatments:
    * No epidural injections or nerve block proc
Time Frame: Baseline and 24 months
Measure: Number; unit: percentage of subjects
Arm/Group | 1 - Study Treatment | 2 - Active Control Treatment
Number analyzed (Participants) | 183 | 187
percentage of subjects | 52.7 | 50.2

ADVERSE EVENTS:
Time Frame: 60 Months
Arm/Group | 1 - Study Treatment | 2 - Active Control Treatment
All-Cause Mortality (participants affected / at risk) | 7/190 | 6/201
Serious Adverse Events (participants affected / at risk) | 113/190 | 117/201
Other Adverse Events (participants affected / at risk) | 82/190 | 100/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 - Study Treatment (N=190) | 2 - Active Control Treatment (N=201)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Allergic Reaction (Immune system disorders) | 2 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Angina (Cardiac disorders) | 2 (2) | 0 (0)
Cerebrovascular Accident (CVA) (Nervous system disorders) | 2 (2) | 1 (1)
Coronary Episode, Ischemic (Cardiac disorders) | 0 (0) | 2 (5)
Deep Infection at the Operative Site (Infections and infestations) | 0 (0) | 2 (3)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dural Leak (Nervous system disorders) | 6 (6) | 2 (2)
Dyspnea (Cardiac disorders) | 0 (0) | 1 (1)
Edema (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 2 (2)
Gastrointestional Bleed (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (2)
Infection (Infections and infestations) | 2 (2) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 5 (5) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Neurological Disorder (Nervous system disorders) | 3 (3) | 3 (3)
Other (General disorders) | 37 (48) | 30 (38) — Other Adverse Events include events not fitting an existing adverse event category, including insomnia, psychological disorder, weight loss, general weakness, ganglion cysts, and drug withdrawal
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 14 (14)
Pain - Buttock or Groin (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
Pneumonia (Infections and infestations) | 6 (7) | 2 (2)
Presence of Osteophyte Formation associated with Severe Disc or Facet Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 3 (3) | 1 (1)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Soft Tissue Damage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Stenosis Symptoms at Index Level (Musculoskeletal and connective tissue disorders) | 22 (23) | 18 (19)
Spinous Process Fracture (Injury, poisoning and procedural complications) | 10 (11) | 5 (5)
Stroke (Nervous system disorders) | 4 (4) | 0 (0)
Transient Ischemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Vertebral Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound Dehiscence or Delayed Healing (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound Drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gallstones (Hepatobiliary disorders) | 0 (0) | 1 (1)
Injury, accidental (Injury, poisoning and procedural complications) | 4 (5) | 4 (4)
Leg pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 13 (14)
Loss of bowel control (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adjacent level degenerative disk disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adjacent level stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Cancer/neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 6 (6)
Cardiovascular (Cardiac disorders) | 7 (9) | 7 (9)
Device dislodgement (General disorders) | 0 (0) | 2 (2)
Device migration (General disorders) | 1 (1) | 3 (4)
Device subsidence (General disorders) | 1 (1) | 0 (0)
Genitiurinary (General disorders) | 8 (8) | 4 (4)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 11 (12) | 19 (21)
Pain - buttock (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 4 (4) | 3 (3)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 - Study Treatment (N=190) | 2 - Active Control Treatment (N=201)
Cancer/Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (13) | 13 (14)
Cardiovascular (Cardiac disorders) | 20 (25) | 16 (20)
Endocrine/Metabolic (Endocrine disorders) | 11 (11) | 11 (13)
Genitourinary (General disorders) | 22 (25) | 17 (17)
Infection (Infections and infestations) | 14 (15) | 16 (17)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 78 (108) | 70 (100)
Neurological Disorder (Nervous system disorders) | 22 (27) | 13 (13)
Other (General disorders) | 14 (15) | 5 (10) — Other Adverse Events including events not fitting a specific adverse event category, including insomnia, psychological disorder, weight loss, general weakness, ganglion cysts, and drug withdrawal
Pain - Back (Musculoskeletal and connective tissue disorders) | 50 (56) | 66 (71)
Pain - Buttock and Groin (Musculoskeletal and connective tissue disorders) | 21 (23) | 13 (13)
Pain - Leg (Musculoskeletal and connective tissue disorders) | 37 (41) | 47 (54)
Spinal Stenosis at Index Level (Musculoskeletal and connective tissue disorders) | 35 (37) | 34 (38)
Spinal Process Fracture (Musculoskeletal and connective tissue disorders) | 22 (24) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT00692276/Prot_SAP_000.pdf